CLINICAL TRIAL: NCT02388698
Title: FDG-PET and Circulating HPV in Patients With Cervical Cancer Treated With Definitive Chemoradiation
Brief Title: FDG-PET and Circulating HPV in Patients With Cervical Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Principal Investigator, Dr. Eric Leung, Radiation Oncologist, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HPVDNA01
Record Dates: First submitted 2015-02-24; First posted 2015-03-17 (Estimated); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Cervical Cancer
Keywords: HPV DNA; PET-CT; Recurrent cervical cancer; chemoradiation
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cervical Swab, PET-CT and plasma HPV (Experimental): Participants will have a cervical swab, and plasma HPV at baseline. In addition, a plasma HPV test drawn after completion of radiation. 3 months post chemoradiation, patients will have a PET-CT and plasma HPV completed. Plasma HPV will be drawn at progression/recurrence, if applicable.
  Interventions: Procedure: Cervical swab; Radiation: PET-CT; Biological: Plasma HPV

INTERVENTIONS:
Procedure: Cervical swab — Cervical Swab at baseline.
  HPV testing at recurrence, if applicable.
Radiation: PET-CT — PET-CT will be completed 3 month post chemoradiation.
Biological: Plasma HPV — Plasma HPV will be drawn at baseline, post radiation, 3 month post chemoradiation and at progression (if necessary).

SUMMARY:
The addition of concurrent chemotherapy to definitive radiation has improved the 5-year survival of women with locally advanced cervical cancer to 58%. To determine if plasma HPV DNA predates clinical recurrence and/or improves the accuracy of metabolic response on FDG-PET at 3 months post completion of radical chemo-radiation in patients with locally advanced cervical cancer. Post therapy FDG-PET can help predict progression free survival and overall survival. In addition plasma HPV can be used to monitor response and detect early recurrence. Prospective study will recruit 20 patients with locally advanced cervical cancer to determine if plasma HPV DNA predates clinical recurrence and/or improves the accuracy response on post-therapy FDG-PET scan at 3 months.

DETAILED DESCRIPTION:
The addition of concurrent chemotherapy to definitive radiation has improved the 5-year survival of women with locally advanced cervical cancer to 58%, there is much room for improvement. Post-therapy FDG-PET at 3 months can help predict progression-free and overall survival. Tumors continually shed their DNA into the circulation, where it can be accessed to measure disease burden. Cervical cancer is caused by Human Papilloma Virus (HPV); plasma HPV DNA could be used to monitor response and detect recurrence early. While plasma HPV DNA has been shown to correlate with prognosis and predict recurrence in other cancers, there is limited data in locally advanced cervical cancer.

This prospective multi-institutional study will recruit 20 patients with locally advanced cervical cancer to determine if plasma HPV DNA predates clinical recurrence and/or improves the accuracy response on post-therapy FDG-PET scan at 3 months. Patients will undergo phlebotomy at the following time-points for the measurement of circulating HPV DNA levels: a) baseline; b) end of radiotherapy;c) 3 months post completion of chemoradiation, along with 3-month FDG-PET and d) at recurrence. This study will provide preliminary estimates of the correlation between plasma HPV DNA level, PET finding and clinical outcome, and inform sample size calculation for a larger study. If proven useful in the future, plasma HPV DNA could enable the identification of patients at high risk of recurrence and individualized treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell carcinoma, adenocarcinoma or adenosquamous carcinoma of the cervix, FIGO stage IB-IVA
* planned for radical radiotherapy and concurrent cisplatin chemotherapy.
* Age ≥ 18 years.
* Life expectancy of greater than 3 months.

Exclusion Criteria:

* Evidence of distant metastases (suspicious paraaortic nodes below the renal vessels allowed if they will be encompassed within the radiation field)
* Patients who have received any anticancer treatment for their cervical cancer.
* Eastern Cooperative Oncology Group (ECOG) performance status > 2
* Other cervical cancer tumor histologies (e.g. small cell, serous)
* Contraindications to 18FDG PET-CT
* Inability to lie supine for radiation and/or 18FDG PET-CT
* Contraindication to radiotherapy (e.g. severe Crohn's disease)
* Contraindication to chemotherapy (e.g. non-reversible renal failure)
* History of another invasive malignancy, except for non-melanoma skin cancer or tumors curatively treated with no evidence of disease for ≥ 5 years.
* Known pregnancy or lactating

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-11-23 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in plasma HPV DNA to 3 months. | Pre treatment and within the first 3 months post treatment
  To determine if HPV DNA predates clinical recurrence and/or improves the accuracy of metabolic response on FDG-PET scan at 3 months post completion of radical chemoradiation in patients with locally advanced cervical cancer

CONTACTS AND LOCATIONS:
Overall Officials: Eric Leung, MD, Principal Investigator — Sunnybrook Research Institute
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada